CLINICAL TRIAL: NCT01019369
Title: Randomized Clinical Trial of Self Versus Clinical Administration of Depot Medroxyprogesterone Acetate
Brief Title: Study of Self or Clinic Administration of DepoProvera
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carolyn L. Westhoff (Other)
Collaborators: Family Planning Fellowship (Other); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Carolyn L. Westhoff, Professor of Obstetrics and Gynecology, Population and Family Health and Epidemiology, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAD8306
Record Dates: First submitted 2009-11-18; First posted 2009-11-25 (Estimated); Results first posted 2015-04-15 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Contraception
Keywords: Contraception; Medroxyprogesterone 17-acetate; Self administration
MeSH Terms: interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self Administration of DMPA (Experimental): Self administration of subcutaneous depot medroxyprogesterone acetate
  Interventions: Drug: Medroxyprogesterone 17-Acetate
- Clinic administration of DMPA (Active Comparator): Clinic administration (routine care) of DMPA
  Interventions: Drug: Medroxyprogesterone 17-Acetate

INTERVENTIONS:
Drug: Medroxyprogesterone 17-Acetate — Depot medroxyprogesterone acetate, SC, every 12 weeks for 1 year
  Other Names: depo-subQ 104
  Arms: Self Administration of DMPA
Drug: Medroxyprogesterone 17-Acetate — Depot medroxyprogesterone acetate, SC, every 12 weeks for 1 year
  Other Names: depo-subQ 104
  Arms: Clinic administration of DMPA

SUMMARY:
Depot medroxyprogesterone acetate (DepoProvera) is an acceptable form of contraception for many women. However, difficulty in access may cause many women to discontinue use, often without the use of another effective method of contraception, thereby leaving them vulnerable to unintended pregnancy. This study will randomly assign women who present for contraceptive services to two groups: self or clinic administered SC DMPA. The participants will be followed for one year to compare continuation rates, acceptability, cost effectiveness, evidence of skin changes, and need for continued support between the two groups.

DETAILED DESCRIPTION:
Unintended pregnancy remains a worldwide problem in both developed and developing countries. In 2001, 49% of pregnancies in the United States were unintended. Moreover, more than 6 million women annually are at high risk of becoming unintentionally pregnant because of a gap in contraceptive use, and disadvantaged women are more likely to have more difficulty than others with continuous method use. Multiple strategies have been explored and implemented to increase the effective usage of contraception, including promoting the use of longer acting reversible contraceptives.

Difficulty in access to depot medroxyprogesterone acetate (DMPA) remains a problem. With the advent of a subcutaneous formulation of DMPA, administration outside of the clinical setting is possible. The acceptability of self administered DMPA has also been reviewed, with favorable outcomes; however, the actual intervention has not been studied.

This study will recruit women presenting for abortion or contraceptive services at the Columbia University and New York Presbyterian affiliated Family Planning Clinic and Special Gynecology Services who desire DMPA for contraception. Women will be randomized to two groups: self administration of SC DMPA or clinic administration of SC DMPA. The primary objective of this study is to compare the continuation rates of SC DMPA between the self and clinic administration groups at 6 months. Secondary outcomes include participant satisfaction, cost effectiveness of self-injected use of DMPA, baseline predictors of method continuation or discontinuation, evidence of persistent skin changes following administration of SC DMPA, and need for continued clinical support.

ELIGIBILITY:
Inclusion Criteria:

1. age greater than or equal to 18 years
2. seeking DMPA for contraception
3. English or Spanish speaking
4. consistent access to a working telephone
5. availability for follow up for one year

Exclusion Criteria:

1. suspected or continuing pregnancy
2. undiagnosed vaginal bleeding
3. known or suspected breast cancer
4. acute liver disease
5. known hypersensitivity to medroxyprogesterone acetate or any other components of DMPA
6. desire for pregnancy within one year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Westhoff, MD, MSc, Principal Investigator — Columbia University; Anitra Beasley, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University/New York Presbyterian Hospital, New York, New York, United States

REFERENCES:
- [Derived] Beasley A, White KO, Cremers S, Westhoff C. Randomized clinical trial of self versus clinical administration of subcutaneous depot medroxyprogesterone acetate. Contraception. 2014 May;89(5):352-6. doi: 10.1016/j.contraception.2014.01.026. Epub 2014 Feb 7. PMID 24656555

RESULTS

PARTICIPANT FLOW:
Groups:
- Self Administration of DMPA: Self administration of subcutaneous (SC) DMPA (depot medroxyprogesterone acetate)
  Medroxyprogesterone 17-Acetate: Depot medroxyprogesterone acetate, SC, every 12 weeks for 1 year
Period: Overall Study
Arm/Group | Self Administration of DMPA | Clinic Administration of DMPA
Started | 86 | 46
Completed | 76 | 39
Not Completed | 10 | 7
Not completed — Lost to Follow-up | 10 | 6
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self Administration of DMPA | Clinic Administration of DMPA | Total
Number analyzed (Participants) | 86 | 46 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (6.1) | 26.1 (6.3) | 26.03 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 46 | 132
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 86 | 46 | 132

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Continuing DMPA at 6 Months
Description: The study was designed to examine if increasing accessibility to DMPA by decreasing the need for multiple clinic visits will increase participant continuation of DMPA
Time Frame: 6 months
Population: Data was analyzed with the assumption that participants who were "lost to follow-up" had discontinued DMPA use.
Measure: Number; unit: participants
Arm/Group | Self Administration of DMPA | Clinic Administration of DMPA
Number analyzed (Participants) | 86 | 45
participants | 61 | 29

2. Secondary Outcome: Number of Participants Continuing DMPA
Description: The study was designed to examine the increasing accessibility to DMPA by decreasing the need for multiple clinic visits will increase method continuation rates at all other endpoints.
Time Frame: 3, 9, 12 months
Population: 115 women w 12 month follow-up data (76 and 39) . 10 participants LTFU in self-administration group, and 7 participants LTFU in the clinic administration group.
Measure: Count of Participants; unit: Participants
Arm/Group | Self Administration of DMPA | Clinic Administration of DMPA
Number analyzed (Participants) | 76 | 39
Participants | 61 | 29

3. Secondary Outcome: Number of Participants Who Would Continue With Self Administration of SC DMPA if it Were Available
Description: The study was designed to examine if self administration of SC DMPA is an acceptable alternative to clinic administration of SC DMPA
Time Frame: 6, 12 months
Population: Data were not collected. No analysis was performed.
Arm/Group | Self Administration of DMPA | Clinic Administration of DMPA
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Prevalence of Participants With Persistent Skin Changes
Description: The study was designed to examine if using SC DMPA will cause skin changes (dimpling, induration, or atrophy)
Time Frame: 12 months
Population: Data were not collected. No analysis was performed.
Arm/Group | Self Administration of DMPA | Clinic Administration of DMPA
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Scaled Satisfaction Score
Description: This study was designed to examine if age, parity, partner support, and personal motivation to avoid pregnancy will predict method continuation rates with questionnaires.
Time Frame: 6, 12 months
Population: Data were not collected. No analysis was performed.
Arm/Group | Self Administration of DMPA | Clinic Administration of DMPA
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Average Minutes Spent Getting Ready for and Giving the Injection
Description: In total, how much time did the participant spend getting ready for and giving the injection. This includes the time the participant spent getting ready to come to the clinic, getting to the appointment, and waiting for the provider for the control group.
Time Frame: 0-12 months
Population: Data were not collected. No analysis was performed.
Arm/Group | Self Administration of DMPA | Clinic Administration of DMPA
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Self Administration of DMPA | Clinic Administration of DMPA
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/46
Other Adverse Events (participants affected / at risk) | 0/86 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No